CLINICAL TRIAL: NCT03429374
Title: Tacks Versus Glue for Mesh Fixation in Laparoscopic Ventral Hernia Repair Treating Defects Between 2 and 5 cm Width: a Multicenter Randomized Controlled Study
Brief Title: Tacks Versus Glue for Mesh Fixation in Laparoscopic Ventral Hernia Repair Treating Defects Between 2 and 5 cm Width
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Limited patient enrollment
Sponsor: Duomed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BLITS-01
Record Dates: First submitted 2018-01-09; First posted 2018-02-12 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Ventral Hernia
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Intervention Model Description: Patients are randomly allocated to group 1 or group 2:
  * Group 1: Mesh fixation with tacks.
  * Group 2: Mesh fixation with glue.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liquiband Fix8 glue mesh fixation (Active Comparator)
  Interventions: Device: Liquiband Fix8
- Mesh fixation with absorbable tacks (Active Comparator)
  Interventions: Device: Absorbable tack

INTERVENTIONS:
Device: Liquiband Fix8 — LiquiBand® Fix 8™ (Advanced Medical Solutions - Plymouth, UK) is a hernia mesh fixation device providing strong and secure mesh fixation without causing any tissue damage or mechanical trauma. This device is designed to offer precise and controlled delivery of tissue glue (n-butyl-2-cyanoacrylate), resulting in a strong mesh fixation.
  Arms: Liquiband Fix8 glue mesh fixation
Device: Absorbable tack — Absorbable tack
  Arms: Mesh fixation with absorbable tacks

SUMMARY:
In laparoscopic ventral hernia repair, an abundance of methods has been developed to fix the mesh to the abdominal wall, including sutures (non-absorbable or absorbable), staples (non-absorbable or absorbable), clips, tacks (non-absorbable or absorbable) and (fibrin and synthetic) glues. Which fixation technique is superior, is still under evaluation. There is clearly a need for larger trials to obtain confident results on the safety and performance of glue mesh fixation and tack mesh fixation in LVHR. The hypothesis of this prospective, randomized controlled study is that post-operative pain at 4 to 6 weeks after mesh fixation with glue (LiquiBand® Fix 8™) will not differ compared to treatment with absorbable tacks during LVHR. A total of 510 patients will be recruited for this trial. This study will assess: pain, hernia recurrence, safety, procedural characteristics, technical success, analgesic intake, period to return to normal activity and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with ventral hernia (primary or incisional) with a defect size between 2 and 5 cm and eligible for laparoscopic repair.
2. Patients with ASA grade I to III.
3. Patient is at least 18 years old.
4. Patient must sign and date the informed consent form prior to treatment.

Exclusion Criteria:

1. Patient with a recurrence of a previously treated ventral hernia repaired with mesh. Recurrences are only allowed to be included after former primary (suture) repair or retromuscular/onlay mesh repair.
2. Patient is treated by open surgery.
3. Patient has more than one defect. Treatment of Swiss-cheese defects (multiple small defects) is allowed if all defects can be treated with one mesh. Total width cannot exceed 5 cm.
4. Patient with a complex hernia, likely not eligible for laparoscopic repair. Complexity is determined by the investigator (adhesions, small bowel resection, etc).
5. Patient with a life expectancy of less than 2 years.
6. Patient is suspected of being unable to comply with the study protocol.
7. Patient with severe chronic obstructive pulmonary disease.
8. Patient with ASA IV or V.
9. Patient is pregnant.
10. Patient needs acute surgery.
11. Patient is scheduled for surgery within 6 weeks after the index-procedure.
12. Patient has fibromyalgia.
13. Patient with depression as shown in patient medical record.
14. Patient is enrolled in another study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-05-20 (Actual)

PRIMARY OUTCOMES:
Pain in both groups at 4-6 weeks after LVHR using the Visual Analog Scale (VAS) | At 4 - 6 weeks
  The VAS scale contains a 0 - 100 grading with 0 equaling no pain and 100 equaling the worst conceivable pain. The patient is asked to select the number on the scale that corresponds to the worst level of pain he/she experiences. Pain is classified into mild (1 - 30 mm), moderate (31 - 60 mm) and severe (61 - 100 mm). Absence of pain is defined as VAS = 0.

SECONDARY OUTCOMES:
Period of hospitalization | up to 5 days
  Record the number of days in hospital until discharge
Operating time | Intra-operatively
Intra-operative adverse events | Intra-operatively
  Intra-operative adverse events include bleeding and enterotomy
Post-operative adverse events | up to 24 months follow-up
  Post-operative adverse events include seroma (i.e. accumulation of wound fluid), ileus (i.e. bowel obstruction), infection, bowel injury, major bleeding requiring blood transfusion or re-intervention, complications due to anesthesia and minor bleeding at a trocar insertion site
Usability of the glue during the index-procedure | Intra-operatively
  Usability scoring: 1 = bad -> 3 = moderate -> 5 = excellent
Technical success of glue fixation | Intra-operatively
  During the index-procedure, the investigator will register whether fixation of the mesh with glue achieved technical success or not. Technical success is defined as successful hernia repair as intended.
Technical success of tack fixation | Intra-operatively
  During the index-procedure, the investigator will register whether fixation of the mesh with tacks achieved technical success or not. Technical success is defined as successful hernia repair as intended.
Pain at baseline using the VAS scale | At baseline
  The VAS scale contains a 0 - 100 grading with 0 equaling no pain and 100 equaling the worst conceivable pain.
Pain at discharge using the VAS scale | Up to 5 days
  The VAS scale contains a 0 - 100 grading with 0 equaling no pain and 100 equaling the worst conceivable pain.
Pain at 12 months follow-up using the VAS scale | At 12 months follow-up
  The VAS scale contains a 0 - 100 grading with 0 equaling no pain and 100 equaling the worst conceivable pain.
Pain at 24 months follow-up using the VAS scale | At 24 months follow-up
  The VAS scale contains a 0 - 100 grading with 0 equaling no pain and 100 equaling the worst conceivable pain.
Postoperative analgesic intake | Up to 24 months follow-up
  Period of intake
Postoperative analgesic intake | Up to 24 months follow-up
  Type of intake
Period to return to normal activity | At 4 - 6 weeks follow-up
  Number of days after the index-procedure at which the patient resumes normal activities.
Quality of life at baseline. | At baseline
  The Carolinas Comfort Scale questionnaire is a validated, disease-specific, quality of life questionnaire developed for patients undergoing hernia repair with mesh. It is a 23-item questionnaire that measures severity of pain, sensation, and movement limitations from the mesh in eight categories. The CCS score is derived by adding the scores from each of the 23 items. The best possible score is 0 and the worst possible score is 115.
Quality of life at 4-6 weeks. | At 4 - 6 weeks follow-up
  CCS questionnaire
Quality of life at 12 months follow-up. | At 12 months follow-up
  CCS questionnaire
Quality of life at 24 months follow-up. | At 24 months follow-up
  CCS questionnaire
Recurrences during follow-up | up to 24 months follow-up
  A clinical examination is conducted to evaluate recurrence. If there is any suspicion of recurrence, an ultrasound or MRI is performed according to hospital practice to distinguish true recurrences from bulging.

CONTACTS AND LOCATIONS:
Locations (11):
- Belgium (11):
  - Hospital Network Antwerp (ZNA) Jan Palfijn, Antwerp
  - General Hospital Sint Jan Brugge, Bruges
  - University Hospital Brussels, Brussels
  - CHU Charleroi, Charleroi
  - General Hospital Sint Vincentius Deinze, Deinze
  - ZOL Genk, Genk
  - University Hospital Leuven, Leuven
  - CHR Namur, Namur
  - General Hospital Nikolaas, Sint-Niklaas
  - Regional Hospital HH Tienen, Tienen
  - General Hospital Delta Torhout, Torhout

IPD SHARING:
Plan to Share IPD: No